CLINICAL TRIAL: NCT04569721
Title: Percutaneous CT-guided Cryoablation of the Splanchnic Nerves for the Management of Type 2 Diabetes
Brief Title: Percutaneous CT-guided Cryoablation of the Splanchnic Nerves
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There was only one subject consented and it was a screen failure. No participants enrolled and study is being closed due to lack of enrollment.
Sponsor: Emory University (Other)
Collaborators: Georgia Research Alliance (Other)
Responsible Party: Principal Investigator, John Prologo, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000619
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CT guided splanchnic cryoablation (Experimental): Obese patients with type 2 diabetes receiving CT guided splanchnic cryoablation.
  Interventions: Device: CT Guided Splanchnic Cryoablation

INTERVENTIONS:
Device: CT Guided Splanchnic Cryoablation — The patient will be sedated and continuously monitored by the anesthesia team, who will be present for the entire procedure. The puncture site will be anesthetized with 1% Lidocaine infiltration. Following tract anesthesia, and utilizing fluoroscopic CT guidance, four cryoablation probes (Ice Rods®) will be advanced, 2 on each side. In addition, a temperature monitoring probe (Boston Scientific, Multipoint 1.5 Thermal Sensor®) will be advanced on each side. The cryoablation process will include a 10-minute freeze, followed by a 3-minute passive thaw, and a brief active thaw to facilitate probe removal. A final scan will be obtained following removal of the probes. After the procedure, a sterile dressing will be applied, and subjects will be monitored for at least 12 hours in an observation bed in the hospital post-procedure.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of freezing (cryoablation) of the splanchnic nerve for management of diabetes. The splanchnic nerves carry signals from the brain to help regulate the way organs function. Quieting these signals, by freezing the splanchnic nerves, may help the body regulate blood sugar. The study procedure will take about 30 minutes and the researchers hope that it will help people to control their blood sugars, lose weight, and possibly improve blood pressure.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a disease of pandemic proportion, affecting approximately 425 million adults worldwide. The incidence of T2D is increasing in most countries and it is predicted that by the year 2045, 629 million adults will be diagnosed with T2D worldwide. Chronically elevated sympathetic activity has been shown to contribute to the development of metabolic syndrome and T2D. Overweight/obese individuals demonstrate elevated noradrenaline and metabolite levels relative to lean healthy individuals - this is particularly concerning since long term prospective studies have shown that noradrenaline levels predict future risk of T2D. Furthermore, dysfunctional sympathetic response to glucose loads is demonstrated amongst those with T2D compared to pre-diabetes. Since the greater splanchnic nerve is the main source of sympathetic input to the viscera, the researchers postulate that denervation of the splanchnic nerve would lead to decreased sympathetic tone, thereby improving glycemic control in patients with T2D. To the researchers' knowledge, this would be the first study to evaluate the role of splanchnic cryoablation as a potential therapeutic for T2D and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes mellitus (T2DM) for <10 years
* HbA1c between ≥7.5% and ≤10.5%
* Willing to comply with study requirements
* Subjects have failed lifestyle interventions as a first line treatment
* Body mass index (BMI) between 30 and 37

Exclusion Criteria:

* Diagnosis of type 1 diabetes or history of diabetic ketoacidosis
* Thyroid disease unless on stable medications for >3 months
* Systemic steroid use within 30 days
* Use of prescription or over the counter weight loss medications within 6 months prior to randomization
* Any condition or major illness that places the subject at undue risk by participating in the study
* Psychiatric condition rendering the subject unable to understand the possible consequences of the study
* Inability to provide informed consent
* Positive pregnancy test at time of cryoablation procedure
* Female subjects who have been pregnant within 6 months or breast-feeding at time of enrollment into the study, or women who plan to become pregnant within the next 12 months
* Diagnosis of anemia, red blood cell (RBC) transfusion in the preceding 3 months or expectation to receive transfusion within the next 12 months, or hemoglobinopathies that would affect HbA1c reliability
* Active or recent infection
* Immunosuppression
* History of coagulopathy or high risk for development of deep vein thrombosis (including congestive heart failure, those who are non-ambulatory, active leukemia/lymphoma, prior thrombotic events, family history of thrombosis)
* History of autonomic dysfunction, including amyloidosis, Parkinson's disease, autoimmune disease, spinal cord injury
* History of heart failure
* History of macro-occlusive vascular disease
* Glomerular filtration rate (GFR) < 60 mL/min/1.73 m2
* History of abnormal pulmonary function or pulmonary intervention (e.g., thoracotomy, thoracentesis, pneumothorax, or thoracic trauma)
* History of or current substance abuse
* Weight gain or loss of >5% during the six months preceding enrollment
* Use of any antihyperglycemic agents aside from metformin or sulfonylurea therapy

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | Month 12
  The number of participant deaths will be used to assess the safety of the study procedure.
Number of Procedure Related Complications | Month 12
  Safety will be assessed by examining procedure related complications, such as bleeding, infection, hypotension, pain, cardiac abnormalities, gastrointestinal abnormalities, or endocrine abnormalities.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline, Months 1, 3, 6, and 12
  HbA1c is a measurement of a persons average blood sugar levels over the prior 3 months. A normal value is below 5.7%. Prediabetes is indicated for levels between 5.7% and 6.4%. Diabetes is diagnosed for values of 6.5% and above.
Change in Fasting Glucose | Baseline, Day 7, Months 1, 3, 6, and 12
  Fasting plasma glucose measures glucose levels after one has fasted for at least 8 hours. Normal values are below 100 mg/dl. Prediabetes is indicated with values between 100 mg/dl and 125 mg/dl. Diabetes is diagnosed when values are at 126 mg/dl and greater.
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, Months 1, 3, 6, and 12
  HOMA-IR is a measure of insulin resistance and is calculated as insulin (uIU/mL) times glucose (mg/dL), divided by 405. Values under 1.0 indicate optimal insulin sensitivity. Values greater than 1.9 indicate early insulin resistance while values over 2.9 indicate significant insulin resistance.
Change in Body Weight | Baseline, Months 1, 3, 6, and 12
  Body weight will be measured in kilograms (kg).
Change in Waist Circumference | Baseline, Months 1, 3, 6, and 12
  Waist circumference will be measured in centimeters (cm).
Change in Waist-to-Hip Ratio | Baseline, Months 1, 3, 6, and 12
  The waist-to-hip ratio is calculated as waist circumference (cm) divided by hip circumference (cm). A healthy ratio for women is 0.85 or less and a healthy ratio for men is 0.9 or less. Ratios of 1.0 and greater are associated with increased risk for illnesses that are associated with being overweight.
Change in Total Cholesterol | Baseline, Months 1, 3, 6, and 12
  Measuring cholesterol is a diagnostic tool used for estimating risk of cardiac disease. Total cholesterol levels below 200 mg/dL are considered normal.
Change in Low-Density Lipoprotein (LDL) | Baseline, Months 1, 3, 6, and 12
  High levels of LDL leads to arteriosclerosis. LDL levels below 100 mg/dL are considered optimal, however, persons with diabetes or cardiac disease are advised to keep levels below 70 mg/dL.
Change in High-Density Lipoproteins (HDL) | Baseline, Months 1, 3, 6, and 12
  HDL values between 40 and 59 mg/dL are considered normal. HDL values under 40 mg/dL are associated with increased risk of developing heart disease and stroke.
Change in Triglyceride Levels | Baseline, Months 1, 3, 6, and 12
  Triglycerides levels measure fat in blood and high triglyceride levels are associated with health concerns such as high blood pressure and diabetes. Normal levels are below 150 mg/dL, borderline high levels are between 150 and 199 mg/dL, and high levels of triglycerides are values of 200 mg/dL and above.
Change in Systolic Blood Pressure | Baseline, Day 7, Months 1, 3, 6, and 12
  Blood pressure is the pressure of circulating blood on the walls of blood vessels, and it is measured in mm Hg. Systolic blood pressure values of less than 120 mm Hg are considered within the normal range.
Change in Diastolic Blood Pressure | Baseline, Day 7, Months 1, 3, 6, and 12
  Blood pressure is the pressure of circulating blood on the walls of blood vessels, and it is measured in mm Hg. Diastolic blood pressure numbers of less than 80 mm Hg are considered within the normal range.
Change in Orthostatic Blood Pressure | Baseline, Day 7, Months 1, 3, 6, and 12
  Blood pressure is obtained while the participant is seated or supine, then the measurement is repeated with the participant standing. Orthostatic hypotension is indicated if systolic blood pressure decreases by 20 mmm Hg or if diastolic blood pressure decreases by 10 mm Hg with the standing measurement.
Change in Serum Catecholamine Measurements | Baseline, Months 1, 3, 6, and 12
  Serum catecholamine measurements assess the amount of dopamine, norepinephrine, and epinephrine in blood. Increased catecholamines are found during times of emotional or physical stress.
Change in Glucose Tolerance | Baseline, Months 1, 3, 6, and 12
  Glucose tolerance will be measured by oral glucose tolerance tests. A normal glucose level is below 140 mg/dL.
Change in Fasting Insulin Levels | Baseline, Day 7, Months 1, 3, 6, and 12
  The fasting insulin test is used to diagnose insulin resistance. Normal values for fasting insulin are below 25 milli-international units per liter (mIU/L).
Change in Fasting C-peptide Levels | Baseline, Day 7, Months 1, 3, 6, and 12
  C-peptide levels are used in diagnosing diabetes. Normal values for fasting C-peptide are between 0.5 and 2.0 nanograms per milliliter (ng/mL). Values higher than 2.0 ng/mL can indicate insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: John D Prologo, MD, Principal Investigator — Emory University
Locations (1):
- Emory Johns Creek Hospital, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No